CLINICAL TRIAL: NCT05604690
Title: A Randomized, Double-Blind, Placebo- and OMV-Controlled Phase I Study to Evaluate the Safety, Tolerance, and Immunogenicity of the Avacc 10 Vaccine Administered Intranasally to Healthy Adult Volunteers
Brief Title: Safety and Efficacy of Intranasal Administration of Avacc 10 Vaccine Against COVID-19 in Healthy Volunteers
Acronym: ITV2002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intravacc B.V. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ITV2002
Record Dates: First submitted 2022-09-15; First posted 2022-11-03 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind. The Sponsor, Investigator, Medical Monitor, study personnel, and participants are not to make any effort to determine which study drug therapy is being received. Unblinded pharmacy (or other qualified site) personnel will be used in this study to prepare the study drug. Assigned unblinded clinical staff will be responsible for overseeing treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Arm: Cohort 1 and 2 (Experimental): Subjects will receive 2 doses of Avacc 10 via intranasal application.
  * Cohort 1 will receive a low dose of Avacc 10
  * Cohort 2 will receive a high dose of Avacc 10.
  Dosage Form: Liquid Unit Dose: Investigational product (IP) in Phosphate Buffered Saline Route of Administration: Intranasal Physical Description: Slightly opalescent in glass vial
  Interventions: Biological: Avacc 10
- OMV Arm: Cohort 1 and 2 (Active Comparator): Subjects will receive 2 doses of Outer Membrane Vesicles (OMV) comparator via intranasal application.
  Dosage Form: Liquid Unit Dose: OMV comparator in TRIS/sucrose buffer Route of Administration: Intranasal Physical Description: Slightly opalescent in glass vial
  Interventions: Combination Product: Outer Membrane Vesicles (OMV) : OMV alone in vehicle
- Placebo Are: Cohort 1 and 2 (Placebo Comparator): Subjects will receive 2 doses of placebo via intranasal application. Dosage Form: Liquid Unit Dose: Placebo in TRIS/sucrose buffer Route of Administration: Intranasal Physical Description: Clear, colorless in glass vial
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Avacc 10 — Intranasal application of either low dose or high dose of Covid 19 vaccine.
  Arms: Treatment Arm: Cohort 1 and 2
Combination Product: Outer Membrane Vesicles (OMV) : OMV alone in vehicle — OMV will be administered via intranasal route.
  Arms: OMV Arm: Cohort 1 and 2
Other: Placebo — Placebo will be administered via intranasal route.
  Arms: Placebo Are: Cohort 1 and 2

SUMMARY:
This study is a Phase I, first-in-human (FIH), double-blind, placebo- and OMV-controlled study of Avacc 10 in healthy adult male and female subjects to investigate the safety, tolerability, and immunogenicity of intranasally administered Avacc 10.

DETAILED DESCRIPTION:
This study is a Phase I, first-in-human (FIH), double-blind, placebo- and OMV-controlled study of Avacc 10 in healthy adult male and female subjects to investigate the safety, tolerability, and immunogenicity of intranasally administered Avacc 10.

Approximately 36 subjects are planned to be enrolled across 2 cohorts (n=18 per cohort). Cohort 1 will receive a low dose of Avacc 10 and Cohort 2 will receive a high dose of Avacc 10.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, a participant has to meet all of the following inclusion criteria:

  1. Healthy male or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, a full physical/neurological examination including vital signs (including systolic and diastolic BP, temperature, and PR), a 12-lead ECG, and clinical laboratory tests).
  2. Participant must have received a vaccination against SARS-CoV-2 or have been exposed to SARS-CoV-2 at least ≥ 4 months prior to the first study dose or shown to be sero-positive to IgG by any of the serological tests marketed as EUA and authorized by the FDA.
  3. Negative test for SARS-CoV-2 at first visit (Day 1) prior to dosing.
  4. Females must be non-pregnant and non-lactating and must use an acceptable, highly effective contraception in the case of heterosexual intercourse.
  5. Males must use highly effective contraception in the case of heterosexual intercourse.
  6. BMI between 18.0 to 32.0 kg/m2 , inclusive; and a total body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
  7. Written or electronic informed consent from the patient prior to any study procedures in a manner approved by a HREC.
  8. Willing and able to comply with the scheduled visits, confinement period, treatment plan, laboratory tests, and other trial procedures and requirements.

Exclusion Criteria:

* A participant who meets any of the following exclusion criteria must be excluded from the study:

  1. Evidence or history of medical conditions which are unstable, or under investigations currently, defined as major changes to management/medication or surgery/hospitalization in the last 12 months, including hematological (including clotting disorders), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, and untreated seasonal allergies at time of dosing).
  2. History of clinically significant autoimmune disorder (such as Guillain-Barré syndrome).
  3. History of febrile illness within 14 days prior to the first dose.
  4. Confirmed SARS-CoV-2 infection within the last 4 months prior to study enrollment.
  5. Known exposure to another person with SARS-CoV-2 infection within the last 14 days prior to study enrolment.
  6. Vaccination with a live vaccine within the 4 weeks prior to study enrollment or any non-live vaccination within the 2 weeks prior to study enrollment, or that is planned during study participation.
  7. Vaccination against N. meningitidis (type B).
  8. History of frequent epistaxis (defined as a weekly occurrence, or more frequently).
  9. Evidence of a deviated septum, or other nasal abnormality, which may impede the ability for intranasal administration of any study medication.
  10. History of, or current positive results for, any of the following serological tests: HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbcAb), or hepatitis C antibody (HCVAb).
  11. Malignancy or a history of malignancy in the previous 5 years, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or adequately treated cervical carcinoma-in-situ.
  12. Documented history of alcohol, cocaine, or IV drug abused within 6 months of study enrollment.
  13. Treatment with an IP within 90 days, preceding study enrollment.
  14. Use of prescription and non-prescription intranasal drug within 7 days prior to first dose of intranasal administration and throughout the study, until 1 month after the last intranasal administration.
  15. Screening supine BP ≥ 155 mmHg (systolic) or ≥ 95 mmHg (diastolic), following at least 5 minutes of supine rest. If BP is ≥ 155 mmHg (systolic) or ≥ 95 mmHg (diastolic), the BP should be repeated 2 more times with the subject at supine rest and the average of the 3 BP values should be used to determine the subjects' eligibility.
  16. Screening 12-lead ECG following at least 5 minutes of supine rest demonstrating a Fridericia corrected QT (QTcF) interval ˃ 450 msec (for males) or > 470 msec (for females) or a QRS interval ≥ 120 msec. If QTcF exceeds 450 msec for men or 470 msec for females, or QRS exceeds ≥ 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF (or QRS) values should be used to determine the subjects' eligibility.
  17. Subjects with clinically significant abnormalities (as determined by the Investigator) in clinical laboratory tests at Screening, as assessed by the study-specific clinical laboratory. A single repeat test may be conducted if deemed necessary. Exception may be granted at the discretion of the Investigator where no confounding factors are expected to impact the safety of the subjects or the integrity of the study
  18. Pregnant, lactating, or planning to become pregnant (self or partner) at any time during the study, or 90 days after last intranasal administration.
  19. Blood or plasma donation of approximately 500 mL or more within 90 days prior to the first intranasal administration.
  20. Previous history of intolerance or hypersensitivity to any component of the IP formulation.
  21. Subjects who have previously experienced a Grade 3 or higher AE to receipt of a SARS-CoV-2 vaccination.
  22. Subjects who are investigational site staff members directly involved in the conduct of this study and their family members, site staff otherwise supervised by the Investigator, and participants who are employees of the Sponsor or are agents of the Sponsor.
  23. Any other reason, criteria that may interfere with the interpretation of study results or, in the judgement of the Investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of intranasal administration of Avacc 10 in healthy subjects by incidence of adverse events. | Screening to end of the follow up period; up to 28 days post final administration period
  Adverse Events will be coded using the most current version of the MedDRA®
To evaluate the safety and tolerability of intranasal administration of Avacc 10 in healthy subjects by evaluating serious adverse events. | Screening to end of the follow up period; up to 28 days post final administration period
  Serious Adverse Events will be coded using the most current version of the MedDRA®
To evaluate the safety and tolerability of intranasal administration of Avacc 10 in healthy subjects by incidence of clinically significant laboratory findings | Screening to end of the follow up period; up to 28 days post final administration period
  Clinical laboratory samples will consist of hematology, biochemistry, and urinalysis
To evaluate the safety and tolerability of intranasal administration of Avacc 10 in healthy subjects by incidence of clinically significant ECG findings | Screening to end of the follow up period; up to 28 days post final administration period
  ECG findings will be used for safety analysis.
To evaluate the safety and tolerability of intranasal administration of Avacc 10 in healthy subjects by incidence of clinically significant vital signs | Screening to end of the follow up period; up to 28 days post final administration period
  BP [systolic and diastolic], PR, and temperature will be measured for analysis of vital signs

SECONDARY OUTCOMES:
To evaluate the immunogenic response of intranasal administration of Avacc 10 in healthy subjects. Immunogenicity evaluations will be done via serum analysis for biomarkers representative of an immunogenic response to a SARSCoV-2 vaccine. | At Screening (at least 3 days prior to first administration), at the follow-up visits 2 weeks following each dose (Day 15 [± 1 day] and Day 36 [± 1 day]), and at the follow-up visit 28 days (window 28-35 days) following the second treatment dose
  Assessment will be performed of the association between changes in immunogenicity outcomes of SARS-CoV-2 NAbs in serum, anti-SARS-CoV-2 IgA and IgG in serum. The Immunogenicity Population will be the primary population for immunogenicity endpoints.
To evaluate the immunogenic response of intranasal administration of Avacc 10 in healthy subjects. Immunogenicity evaluations will be done via nasal wash analyses for biomarkers representative of an immunogenic response to a SARS-CoV-2 vaccine. | At Screening (at least 3 days prior to first administration), at the follow-up visits 2 weeks following each dose (Day 15 [± 1 day] and Day 36 [± 1 day]), and at the follow-up visit 28 days (window 28-35 days) following the second treatment dose
  Assessment will be performed of the association between changes in immunogenicity outcomes of anti-SARS-CoV-2 IgA in nasal wash. The Immunogenicity Population will be the primary population for immunogenicity endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Sunshine Coast Clinical Trial Centre, Sippy Downs, Queensland, Australia